CLINICAL TRIAL: NCT05285501
Title: Immersive Virtual Therapeutic Garden as a Support for Late-Life Depressive Symptoms: a Randomized Clinical Trial
Brief Title: Virtual Therapeutic Garden for Depressive Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wroclaw University of Health and Sport Sciences (Other)
Collaborators: Foundation for Senior Citizen Activation SIWY DYM (Other)
Responsible Party: Principal Investigator, Błażej Cieślik, Principal Investigator, Wroclaw University of Health and Sport Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 59/0203/S/05
Record Dates: First submitted 2022-03-08; First posted 2022-03-17 (Actual); Last update posted 2022-09-30 (Actual); Status verified 2022-09

CONDITIONS: Depressive Symptoms; Depression; Anxiety
Keywords: virtual reality; depression; anxiety; mental health; elderly; rehabilitation; virtual garden
MeSH Terms: conditions — Depression; Anxiety Disorders; Psychological Well-Being

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Therapeutic Garden (Experimental): Twice a week, for a 4 consecutive weeks:
  8 sessions of general fitness training (40 minutes each) 8 sessions of VRTierOne therapy (20 minutes each)
  Interventions: Behavioral: Group general fitness training; Device: VRTierOne
- Control (Active Comparator): Twice a week, for a 4 consecutive weeks:
  8 sessions of general fitness training (40 minutes each) 8 sessions of group relaxation and psychoeducation (20 minutes each)
  Interventions: Behavioral: Group general fitness training; Behavioral: Group relaxation and psychoeduaction

INTERVENTIONS:
Behavioral: Group general fitness training — A single session of general fitness training will be composed of low-intensity, general-fitness exercises. Most of the exercises will be carried out in a sitting position and standing positon. The session will contain aerobic (general warm-up), musculo-articular (strengthening muscles and joints range of motion) and stabilizing exercises (improve spatio-visual coordination). Conducted by a physiotherapist in group form.
Behavioral: Group relaxation and psychoeduaction — A single session of relaxation (10 minutes) psychoeducation (10 minutes) will contain minilectures about mental well-being and psychohygiene. In summary 20 minutes.
  Arms: Control
Device: VRTierOne — As a virtual reality source, VRTierOne device (Stolgraf®) were used. Thanks to using head mounted display and the phenomenon of total immersion "VRTierOne" Stolgraf® provides an intense visual, auditory and kinesthetic stimulation. It can have a calming and mood-improving effect or help the patients recognize their psychological resources and motivate to the rehabilitation process. In the virtual therapeutic garden there are a rich set of symbols and metaphors based on Ericksonian Psychotherapy approach. The most important is the Garden of Revival which symbolizes the patient's health. It used to be full of life and energy, now it is neglected, requires work to be revived. In the therapeutic process day by day, the lector (therapist) tells the patient a symbolic story about his/her situation. By performing tasks in the virtual garden, the patient influences the course of this story, becomes an active participant of the therapeutic process and sees the effects his work.
  Arms: Virtual Therapeutic Garden

SUMMARY:
This study evaluates the addition of virtual therapy intervention in the treatment of depression in the elderly. Half of the participants will receive virtual reality treatment as an addition to physical exercises and psychoeducation, while the other half will receive physical exercises and psychoeducation alone.

DETAILED DESCRIPTION:
Depressive disorders are frequent and can either first be manifested at a younger age and recurrent during later life or have an onset beyond 60 years (late-life depression). The multifactorial genesis of depression in old age includes psychosocial, vascular and metabolic factors and requires multimodal and multi-professional therapy including physical activity and psychosocial interventions. However, there is still a percentage of older people who do not show improvement in depressive symptoms.

In recent years, various types of virtual reality are gaining in popularity, primarily because of the availability and ease of use. A systematic review from 2018 concluded that VR treatment had moderate to large effects in anxiety and depression, compared to controls and it could be another effective choice available to clinicians and patients.

Therefore, the aim of this project was to evaluate the effectiveness of virtual therapy in the elderly, in whom the previous multimodal therapeutic program has not brought the expected results.

ELIGIBILITY:
Inclusion Criteria:

* GDS≥10 or HADS-A≥8 or HADS-D≥8

Exclusion Criteria:

* cognitive impairment (MMSE<24);
* aphasia and a serious loss of sight or hearing that makes it impossible to assess cognitive functions based on MMSE;
* contraindications for virtual therapy (epilepsy, vertigo, eyesight impairment);
* substance abuse;
* participation in another therapeutic project or individual psychotherapy;
* antidepressant treatment;

Ages: 60 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-03-15 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
The Geriatric Depression Scale (GDS)(Change from baseline) | 15 minutes
  The Geriatric Depression Scale is a self-report 30-items measure of well-being and mood in older adults. The patient responds in a "Yes/No" format. Scoring ranges from 0 to 30, where 11 and more means mood disorders. The higher score means the greater depression.

SECONDARY OUTCOMES:
Hospital Anxiety and Depression Scale (HADS)(Change from baseline) | 30 minutes
  The Hospital Anxiety and Depression Scale (HADS) is a fourteen-item scale scoring from 0 to 3 for each item. The first seven items relate to anxiety (HADS-A), and the remaining seven items relate to depression (HADS-D). The global scoring ranges from 0 to 42 with a cut-off point of 8/21 for anxiety and 8/21 for depression. The higher the score, the greater anxiety or depression symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Joanna Szczepańska-Gieracha, Professor, Study Director — University School of Physical Education, Wroclaw, Poland; Błażej Ł Cieślik, PhD, Principal Investigator — Jan Dlugosz University in Czestochowa, Poland
Locations (2):
- Poland (2):
  - Foundation for Senior Citizen Activation SIWY DYM, Wroclaw, Lower Silesian Voivodeship
  - University School of Physical Education, Wroclaw, Lower Silesian Voivodeship

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cieslik B, Mazurek J, Rutkowski S, Kiper P, Turolla A, Szczepanska-Gieracha J. Virtual reality in psychiatric disorders: A systematic review of reviews. Complement Ther Med. 2020 Aug;52:102480. doi: 10.1016/j.ctim.2020.102480. Epub 2020 Jun 9. PMID 32951730
- [Background] Jozwik S, Cieslik B, Gajda R, Szczepanska-Gieracha J. The Use of Virtual Therapy in Cardiac Rehabilitation of Female Patients with Heart Disease. Medicina (Kaunas). 2021 Jul 28;57(8):768. doi: 10.3390/medicina57080768. PMID 34440974
- [Background] Szczepanska-Gieracha J, Jozwik S, Cieslik B, Mazurek J, Gajda R. Immersive Virtual Reality Therapy as a Support for Cardiac Rehabilitation: A Pilot Randomized-Controlled Trial. Cyberpsychol Behav Soc Netw. 2021 Aug;24(8):543-549. doi: 10.1089/cyber.2020.0297. Epub 2021 Feb 11. PMID 33577375
- [Background] Szczepanska-Gieracha J, Cieslik B, Serweta A, Klajs K. Virtual Therapeutic Garden: A Promising Method Supporting the Treatment of Depressive Symptoms in Late-Life: A Randomized Pilot Study. J Clin Med. 2021 May 1;10(9):1942. doi: 10.3390/jcm10091942. PMID 34062721
- [Background] Jozwik S, Cieslik B, Gajda R, Szczepanska-Gieracha J. Evaluation of the Impact of Virtual Reality-Enhanced Cardiac Rehabilitation on Depressive and Anxiety Symptoms in Patients with Coronary Artery Disease: A Randomised Controlled Trial. J Clin Med. 2021 May 16;10(10):2148. doi: 10.3390/jcm10102148. PMID 34065625
- [Background] Rutkowski S, Rutkowska A, Kiper P, Jastrzebski D, Racheniuk H, Turolla A, Szczegielniak J, Casaburi R. Virtual Reality Rehabilitation in Patients with Chronic Obstructive Pulmonary Disease: A Randomized Controlled Trial. Int J Chron Obstruct Pulmon Dis. 2020 Jan 13;15:117-124. doi: 10.2147/COPD.S223592. eCollection 2020. PMID 32021150
- [Derived] Cieslik B, Juszko K, Kiper P, Szczepanska-Gieracha J. Immersive virtual reality as support for the mental health of elderly women: a randomized controlled trial. Virtual Real. 2023 May 7:1-9. doi: 10.1007/s10055-023-00797-w. Online ahead of print. PMID 37360811